CLINICAL TRIAL: NCT01353547
Title: Integrating Genetic and Environmental Risk Scores Into an Algorithm to Predict Multiple Sclerosis Susceptibility
Brief Title: Genes and Environment in Multiple Sclerosis
Acronym: GEMS
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: University of Pittsburgh (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Philip De Jager, Professor of Neurology, Columbia University
Other Study IDs: AAAR4456
Record Dates: First submitted 2011-05-11; First posted 2011-05-13 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
Keywords: genomic analysis; online surveys; biological specimen collection
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Sample (required), Blood Sample (optional), Stool Sample (optional) Biospecimen collection is done remotely by mailing kits to subjects. Coded samples are stored at Columbia University Medical Center (CUMC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Received anti-TNFa therapy: Received anti-TNFa therapy
- First-degree relative of MS patients: First-degree relative (child, parent or sibling) of a diagnosed MS patient
  A subgroup will be asked to undergo magnetic resonance imaging (MRI). Participants may be asked to donate a stool sample for gut flora analysis and a blood sample for ribonucleic acid (RNA) sequencing.
- Referred by the Partners MS Center: Referred by the Partners MS Center

SUMMARY:
The purpose of the research study is to identify the genetic, environmental and immune profiles that may increase a person's risk of developing multiple sclerosis (MS). While MS is not a disease caused by a single variation in genetic material (DNA), a single environmental factor, or a single malfunction in immune cells, there are genetic alterations, environmental exposures and immunologic factors that make the development of MS more likely. Obtaining information about who is at risk for MS will be beneficial in the future if the investigators can identify effective ways to prevent or slow down the progression of this disease.

DETAILED DESCRIPTION:
MS is an autoimmune disease in which the immune system (white bloods cells that normally fight infection) becomes misdirected and attacks healthy tissue. In patients with MS, the misdirected white blood cells attack myelin, a lining that insulates the nerves found in the brain and spinal cord. This results in inflammation and damage in the myelin. Loss of this protective lining disrupts nerve impulses and causes abnormal function in the nervous system.

This large research study will ultimately enroll 5000 subjects who are at risk of developing MS.

ELIGIBILITY:
Inclusion Criteria:

* First Degree Relatives of Patients with MS, or
* Patients who have received anti-TNFa therapy as treatment for inflammatory diseases other than MS such as Crohn's disease, psoriasis and rheumatoid arthritis, or
* Patients that have been referred for an evaluation of first presentation of neurologic symptoms but do not have a diagnosis of MS
* Live in the United States

Exclusion Criteria:

* Does not match any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This large research study will ultimately enroll over 10000 subjects who are at risk of developing MS. The study will last 20 years. We will recruit subjects from all over the United States, as everything is done via mail, email, or/and phone.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2040-10 (Estimated); Study Completion 2040-10 (Estimated)

PRIMARY OUTCOMES:
Total number of subjects who are diagnosed with MS | 20 years
  For each subject, weighted integrated risk score will be calculated, combining genetic burden and environmental exposure. A distribution of the risk score will be generated for the cohort. At this stage, the study will assess whether there is an increase in subjects with a diagnosis of MS (validated by a letter or copy of clinical records from the subject's neurologist) within the higher end vs. the lower end of the risk score distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Zongqi Xia, MD, PhD, Study Director — University of Pittsburgh
Locations (5):
- United States (5):
  - National Institute of Neurological Disorders and Stroke, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Columbia University Irving Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia Z, Steele SU, Bakshi A, Clarkson SR, White CC, Schindler MK, Nair G, Dewey BE, Price LR, Ohayon J, Chibnik LB, Cortese IC, De Jager PL, Reich DS. Assessment of Early Evidence of Multiple Sclerosis in a Prospective Study of Asymptomatic High-Risk Family Members. JAMA Neurol. 2017 Mar 1;74(3):293-300. doi: 10.1001/jamaneurol.2016.5056. PMID 28114441